CLINICAL TRIAL: NCT05809726
Title: Does Manual Lymph Drainage Affect Autonomic Functions in Healthy Women?
Brief Title: The Effects of Manual Lymphatic Drainage on the Autonomic Nerve System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/03-06
Record Dates: First submitted 2023-01-25; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: manual lymph drainage; autonomic function; heart rate variability; cold pressure test
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual lymph drainage group (Experimental): Manual lymph drainage; neck drainage, abdominal drainage, stimulation of axillary lymph nodes, and right arm drainage were performed by following a special technique and sequence. MLD was applied in a comfortable position while the patient was lying in the supine position. It took an average of 20 minutes.
  Interventions: Other: Manual lymph drainage
- Sham manual lymph drainage group (Sham Comparator): Sham manual lymph drainage; deep pressure was applied from distal to proximal with rapid movements to the right extremity to which the cold pressure test was applied. Fingers, dorsal and palmar surfaces of the hand, forearm, elbow, and upper arm were applied in order. The application was performed while the patient was lying in the supine position and lasted an average of 20 minutes.
  Interventions: Other: Manual lymph drainage
- Control Group (No Intervention): Participants in the control group were asked to lie on their backs for 10 minutes without speaking in a quiet, calm environment. At the end of 10 minutes, the patient was placed in a sitting position again and the third evaluation was performed.

INTERVENTIONS:
Other: Manual lymph drainage — one session 20 minutes
  Other Names: Sham manual lymph drainage
  Arms: Manual lymph drainage group; Sham manual lymph drainage group

SUMMARY:
Forty healthy women who met the inclusion criteria were included in the study. In the single-blind randomized controlled study, the participants were divided into 3 groups manual lymphatic drainage(MLD), sham MLD, and control group. After evaluating the demographic information, blood pressure, and heart rate variability (HRV) of the participants, the cold pressure test was applied. Immediately after the test, blood pressure and HRV were re-evaluated. The MLD group received short neck, abdominal, and lymph node stimulation and right arm MLD applications. A sham protocol was applied to the sham MLD group. The control group was asked to lie on their back for 10 minutes. After the application, blood pressure and HRV were re-evaluated.

DETAILED DESCRIPTION:
The participants included in the study were randomly divided into 3 groups; manual lymph drainage, sham manual lymph drainage, and a control group in the computer program.

Participants rested for 5 minutes before the first evaluation. The first evaluation was made after the demographic information of the participant was obtained. Within the scope of this evaluation, blood pressure, heart rate, and heart rate variability were evaluated. All assessments were performed on the patient's dominant upper extremity. After the evaluation, cold pressure test was applied to the dominant extremity. A second assessment was made immediately after the test. All of the parameters examined within the scope of the first evaluation were examined for the second time. Appropriate treatment was applied to the group to which the participant belonged. After the treatment, the third evaluation was made and the study was terminated. All participants were asked to avoid exercise, caffeine, energy drinks, and heavy meals at least 1 hour before the test. Environmental noise, light, and temperature were controlled during the test.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years of age
* being voluntary to participate in the study

Exclusion Criteria:

* having advanced cardiorespiratory diseases
* orthopedic and neurological problems
* using medication related to pain
* cardiovascular system, having skin disorders that prevent skin contact
* having cold urticaria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
autonomic functions assessment | 1 year
  heart rate variability
physiological parameter | 1 year
  Systolic blood pressure (mmHg) and diastolic blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim SJ, Kwon OY, Yi CH. Effects of manual lymph drainage on cardiac autonomic tone in healthy subjects. Int J Neurosci. 2009;119(8):1105-17. doi: 10.1080/00207450902834884. PMID 19922342
- [Result] Honguten A, Mekhora K, Pichaiyongwongdee S, Somprasong S. Effects of lymphatic drainage therapy on autonomic nervous system responses in healthy subjects: A single blind randomized controlled trial. J Bodyw Mov Ther. 2021 Jul;27:169-175. doi: 10.1016/j.jbmt.2021.03.019. Epub 2021 Mar 28. PMID 34391230
- [Result] Schingale FJ, Esmer M, Kupeli B, Unal D. Investigation of the Less Known Effects of Manual Lymphatic Drainage: A Narrative Review. Lymphat Res Biol. 2022 Feb;20(1):7-10. doi: 10.1089/lrb.2019.0091. Epub 2021 Mar 22. PMID 33751912